CLINICAL TRIAL: NCT02742805
Title: Sustained Effect of Urticaria Remission With Relatively High Dose Vitamin D Supplementation After Omalizumab Discontinuation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Selina Gierer, D.O. (Other)
Responsible Party: Sponsor-Investigator, Selina Gierer, D.O., Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002729
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Urticaria
Keywords: hives
MeSH Terms: conditions — Urticaria | interventions — Vitamin D; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Vitamin D (Experimental): Participants receive high dose of Vitamin D (4,000 IU/day) in addition to standard of care dose of Omalizumab.
  Interventions: Dietary Supplement: Vitamin D (4,000 IU/day); Drug: Omalizumab
- Low Dose Vitamin D (Active Comparator): Participants receive low dose of Vitamin D (400 IU/day) in addition to standard of care dose of Omalizumab.
  Interventions: Dietary Supplement: Vitamin D (400 IU/day); Drug: Omalizumab

INTERVENTIONS:
Dietary Supplement: Vitamin D (4,000 IU/day) — High Dose of 4,000 IU/day.
  Arms: High Dose Vitamin D
Dietary Supplement: Vitamin D (400 IU/day) — Low Dose of 400 IU/day.
  Arms: Low Dose Vitamin D
Drug: Omalizumab — Standard of care dose.
  Other Names: Xolair

SUMMARY:
The proposed research is intended to determine if supplementation of relatively high dose vitamin D in chronic urticaria patients receiving omalizumab will result in continued symptomatic control of hives after the discontinuation of omalizumab.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed chronic urticaria
* Currently be receiving omalizumab therapy for the treatment of chronic idiopathic urticaria and be well controlled with a USS <25

Exclusion Criteria:

* Not capable of informed consent.
* Not capable of answering the questionnaire.
* Subjects with a pure physical urticaria.
* Pregnant or lactating women.
* Subjects with hypercalcemia (calcium > 10.3 mg/dl) or renal insufficiency (GFR <50 ml/min).
* Subjects with prior anaphylaxis to omalizumab.
* Currently taking high dose vitamin D supplementation.
* Prior high dose vitamin D supplementation for urticaria with failure.
* Baseline 25(OH)D >80 ng/ml
* Subjects with sarcoidosis, hyperparathyroidism, histoplasmosis, lymphoma or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in total Urticaria Severity Score (USS) | Change from Baseline to Month 6
  The USS is a questionnaire which is used to measure urticaria severity. The questionnaire is comprised on 9 questions with each question having 7 total responses on a likert-type scale. Responses to each question range from 0 to 7.

SECONDARY OUTCOMES:
Number of subjects restarted on Omalizumab | 8 Months
  Number of participants restarted on Omalizumab after coming off it at Month 4
Change in total Urticaria Severity Score (USS) | Change from Baseline to Month 8

CONTACTS AND LOCATIONS:
Overall Officials: Selina Gierer, D.O., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States